CLINICAL TRIAL: NCT05010993
Title: Establishing Czech Norms of Selected Standardized Tests for Use in Rehabilitation and Upper Limbs Functional Evaluation
Brief Title: Establishing Czech Norms of Selected Standardized Tests
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kateřina Rybářová, Mgr. Kateřina Rybářová (Master in Occupational Therapy), Charles University, Czech Republic
Other Study IDs: EK-1340.14/20
Record Dates: First submitted 2021-08-12; First posted 2021-08-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Motor Activity
Keywords: standardized test; occupational therapy; fine motor skills; Nine Hole Peg Test; Purdue Pegboard Test; Box and Block Test; Czech language; norms; healthy population
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Czech healthy people: Czech healthy men and women will be asked to fill in a questionnaire. Then they will be tested by the Nine Hole Peg Test, the Purdue Pegboard Test and the Box and Block Test.
  Interventions: Diagnostic Test: Nine Hole Peg Test; Diagnostic Test: Purdue Pegboard Test; Diagnostic Test: Box and Block Test

INTERVENTIONS:
Diagnostic Test: Nine Hole Peg Test — Each person will be tested by the Nine Hole Peg Test (3 attempts per subtest)
Diagnostic Test: Purdue Pegboard Test — Each person will be tested by the Purdue Pegboard Test (3 attempts per subtest)
Diagnostic Test: Box and Block Test — Each person will be tested by the Box and Block Test (3 attempts per subtest)

SUMMARY:
The main aim of the project is to establish Czech updated manuals for the Nine Hole Peg Test, Purdue Pegboard Test and Box and Block Test to be used in rehabilitation to evaluate upper limb functions, including establishing norms for the Czech healthy population.

DETAILED DESCRIPTION:
The main aim of the project is to establish Czech updated manuals for the Nine Hole Peg Test, Purdue Pegboard Test and Box and Block Test to be used in rehabilitation to evaluate upper limb functions, including establishing norms for the Czech healthy population.

The Czech updated manuals for those tests were made by back-translation method and updated for unification of recommended three trials of each subtest administration and interpretation of tested individuals performance.

At least 540 individuals (20-65 years old) will be tested by the updated Czech manuals till the end of 2023 by those three tests. The Czech norms will be established from acquired data.

ELIGIBILITY:
Inclusion Criteria:

* Czech language as a mother tongue
* age from 20 to 65 years

Exclusion Criteria:

* diagnosed pathology of the upper limbs or diseases that negatively affect the dexterity of their limbs
* use of drugs affecting attention
* vision impairment uncorrectable with glasses
* severe hearing loss
* inability to understand instructions
* inability to read or write
* inability to complete testing
* failure to sign Informed consent for probation with inclusion to research and Consent to the collection and processing of personal data during the study at the General University Hospital in Prague

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — based on self-representation
Study Population: Czech healthy men and women
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
results from the Nine Hole Peg Test | 10 minutes
  time in seconds and hundreds of seconds
results from the Purdue Pegboard Test | 25 minutes
  number of parts put in the Pegboard according to the rules
results from the Box and Block Test | 30 minutes
  number of transported blocks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No